CLINICAL TRIAL: NCT05138146
Title: A Single Arm，Open Label，Multi-centers，Phase 2 Study, Aimed to Evaluate the Efficacy and Safety of Recombinant Anti-PD-1 Humanized Monoclonal Antibody Injection (609A) Combined With Doxorubicin Hydrochloride in the Treatment of Metastatic/Unresectable Non-specific Soft Tissue Sarcoma
Brief Title: A Phase 2 Clinical Study of Evaluation of Recombinant Anti-PD-1 Humanized Monoclonal Antibody Injection (609A) Combined With Doxorubicin Hydrochloride in the Treatment of Metastatic/Unresectable Non-specific Soft Tissue Sarcoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sunshine Guojian Pharmaceutical (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SSGJ-609A-ADM-STS-II-01
Record Dates: First submitted 2021-11-14; First posted 2021-11-30 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Sarcoma, Soft Tissue
MeSH Terms: conditions — Sarcoma | interventions — Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental group (Experimental): 609A combined with doxorubicin hydrochloride
  Interventions: Drug: 609A; Drug: doxorubicin hydrochloride

INTERVENTIONS:
Drug: 609A — 609A 200mg,IV, Day 1of each treatment cycle, up to disease progression or intolerable toxicity, death, early withdrawal from the study or loss to follow-up, withdrawal of consent, or the end of the treatment period, whichever occurs first.
  Every 3 weeks a treatment cycle.
Drug: doxorubicin hydrochloride — 60mg/m2 or 75mg/m2, IV, Day1of the1-6th treatment cycles only. Every 3 weeks a treatment cycle.

SUMMARY:
This is a single arm, open label, phase 2 study aimed to evaluate the efficacy and safety of the combination recombinant anti-PD-1 humanized monoclonal antibody injection (609A) and doxorubicin hydrochloride in the treatment of metastatic/unresectable non-specific soft tissue sarcoma

DETAILED DESCRIPTION:
This is a single-arm, open, multi-center phase 2 study aimed at evaluating the efficacy and safety of 609A combined with doxorubicin hydrochloride in patients with metastatic/unresectable non-specified soft tissue sarcoma. This study is divided into the first part (safety introduction period) and the second part (phase II).

Part 1: Security lead-in period The safety lead-in period adopts a single-arm, open design to evaluate the safety, tolerability and preliminary effectiveness of 609A combined with doxorubicin hydrochloride. Which aimed to explore the Recommended phase II dose (RP2D).

Part 2: Phase 2 This part adopts a single-arm, open, Simon two-stage design to further evaluate the anti-tumor efficacy and safety of 609A combined with doxorubicin hydrochloride.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and voluntarily sign an informed consent form;
* Age ≥ 18 years old when signing the informed consent form, regardless of gender;
* Agree to provide biopsy tissue samples or archived tumor tissue samples (part 1 is voluntary);
* Unresectable (including patients who refuse surgical resection) or metastatic unspecified soft tissue sarcoma confirmed by histology/cytology (subtypes allowed to be included include: synovial sarcoma, mucinous/round cell liposarcoma , Uterine leiomyosarcoma, pleomorphic liposarcoma, myxofibrosarcoma, epithelioid sarcoma, pleomorphic rhabdomyosarcoma, leiomyosarcoma, malignant peripheral nerve sheath tumor, angiosarcoma, scalp and facial angiosarcoma, dedifferentiated liposarcoma) patients ；
* Patients who have not received systemic drug therapy in the past;
* According to the RECIST V1.1 solid tumor efficacy evaluation standard, the patient has at least one imaging measurable lesion;
* ECOG score 0 or 1;
* Expected lifetime ≥ 3 months;
* The organ function level must meet the following requirements:

  1. The absolute value of neutrophils (ANC) ≥ 1.5×109/L; platelet count (PLT) ≥100×109/L; hemoglobin (Hb) ≥90 g/L or ≥5.6 mmol/L (not accepted within 14 days) Blood transfusion, albumin or use of EPO, G-CSF);
  2. Total bilirubin (TBIL) ≤ 1.5 × upper limit of normal (ULN), aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) ≤ 2.5 × ULN (for patients with primary liver sarcoma or liver metastases, TBIL is allowed ≤ 3×ULN, AST and/or ALT ≤ 5×ULN), albumin (ALB) ≥ 2.5 mg/dL;
  3. Serum creatinine (Cr) ≤ 1.5×ULN or estimated creatinine clearance (CrCl) ≥ 60 mL/min (Cockroft and Gault formula);
  4. International normalized ratio (INR) ≤ 1.5×ULN; partial activated thromboplastin time (APTT) ≤ 1.5×ULN.
* Female and male patients during the reproductive period need to agree to adequate contraception (such as abstinence, intrauterine device, contraceptives or condoms) during the study period and 6 months after the last dose.

Exclusion Criteria:

* Received radiotherapy covering more than 30% of the bone marrow area or carried out large-area irradiation within 4 weeks before the first administration (palliative radiotherapy for bone or palliative radiotherapy for superficial lesions is allowed, and it has ended 14 days before the first administration );
* Received Chinese medicine or Chinese medicine preparation with anti-tumor as indication within 2 weeks or 5 half-life period (whichever is the elder) before the first administration;
* Those who have participated in and received clinical trials of investigational drugs or interventional devices 4 weeks before the first administration or at least 5 half-lives of the drug (whichever is the elder);
* Vaccination with live attenuated vaccine within 4 weeks before the first administration (seasonal influenza vaccine for injection is generally an inactivated vaccine, which is allowed to be used; while intranasal influenza vaccine [such as flu spray] is a live attenuated vaccine, which is not Allowed)
* Use moderate or strong CYP3A4, P-glycoprotein, CYP2D6 inhibitors and CYP3A4, P-glycoprotein inducers within 1 week before the first administration;
* Any toxicity related to previous radiotherapy has not recovered to ≤ Grade 1 (except for hair loss or treatment-related Grade 2 peripheral neuropathy);
* Patients with active central nervous system (CNS) metastasis and/or cancerous meningitis found in a known or screening phase examination;
* Spinal cord compression that has not been cured by surgery and/or radiotherapy;
* Accompanied by unstable pleural effusion or ascites or pericardial effusion with obvious symptoms (those with stable clinical symptoms after treatment with pleural effusion or ascites or pericardial effusion can be included in the group);
* Those who have a history of other malignant tumors, except for malignant tumors that have undergone radical resection and have not recurred within 5 years after surgery, such as cervical carcinoma in situ and skin basal cell carcinoma;
* Anyone who has been allergic to protein drugs or recombinant proteins or excipients in 609A pharmaceutical preparations in the past;
* People with active tuberculosis (tuberculous bacilli);
* Those who have a history of non-infected pneumonia in the past or who are currently suffering from pneumonia;
* Accompanied by immunodeficiency or active autoimmune disease (in the past 2 years, systemic glucocorticoid systemic treatment with >10 mg/day prednisone or its equivalent is required, but alternative therapies such as thyroxine, Insulin or physiological corticosteroid replacement therapy for adrenal or pituitary insufficiency is not considered a form of systemic therapy and can be admitted to the group), and those who have used any other form of immunosuppressant within 14 days before the first administration ( The use of physiological doses of glucocorticoids can be approved after inquiring the sponsor);
* Those who have received organ or bone marrow transplant in the past;
* Those who have performed or planned to perform major surgery within 28 days before the first medication (except for the operation of establishing vascular access, or performing biopsy through mediastinoscopy or thoracoscopy);
* Actively infected persons who require systemic treatment within 14 days of the first administration;
* Patients with clinically significant cardiovascular and cerebrovascular diseases, including but not limited to:

  1. Congestive heart failure (New York Heart Association classification III-IV);
  2. Poorly controlled hypertension (systolic blood pressure> 160 mmHg and/or diastolic blood pressure> 100 mmHg after treatment with a stable dose of antihypertensive drugs);
  3. Severe arrhythmias that require treatment (except for atrial fibrillation and paroxysmal supraventricular tachycardia);
  4. Myocardial infarction, unstable angina, cerebrovascular accident/stroke occurred within 6 months before the first administration;
  5. Left ventricular ejection fraction (LVEF) of echocardiography <50%;
  6. 3 consecutive 12-ECG average corrected QT intervals (QTcF)> 450 ms (male) or (QTcF)> 470 ms (female) in the resting state;
* Hepatitis B (hepatitis B surface antigen [HbsAg] positive or core antibody [HbcAb] positive and HBV DNA ≥ the lower limit of detection), hepatitis C (hepatitis C virus [HCV] antibody positive and HCV RNA positive), human immunodeficiency People infected with the virus (HIV);
* Those who have abnormal thyroid function tests and are judged by the investigator to be unsuitable to participate in this study;
* Any other serious illness (for example: uncontrolled diabetes, active gastric ulcer, uncontrolled epilepsy, gastrointestinal bleeding, coagulopathy with severe symptoms and signs), mental, psychological, according to the researcher Judging that it may interfere with the planning, treatment and follow-up of the trial, or affect the compliance of the subject, or put the subject at a high risk of treatment-related complications;
* Any other situation in which the investigator judges that the patient is not suitable for entry into this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-12-30 (Estimated); Primary Completion 2023-11-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Recommended phase II dose (RP2D) (Part 1) | At the end of Cycle 2 (each cycle is 21 days)
  RP2D of the combination 609A and doxorubicin hydrochloride.
Adverse events (Part 1) | up to 2 years.
  Evaluate the safety of the combinations According to the National Cancer Institute (NCI) Common Terminology for Adverse Events (CTCAE) .
Objective Response Rate (ORR) (part 2) | Up to 2 years .
  Evaluated per Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT. Complete Response (CR) is a complete elimination of the tumor; Partial Response (PR) is 30% reduction. If a subject experienced a PR, this was required to be confirmed with a second scan at the next appropriate cycle.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) (part 1) | Up to 2 years.
  Evaluated per Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT. Complete Response (CR) is a complete elimination of the tumor; Partial Response (PR) is 30% reduction. If a subject experienced a PR, this was required to be confirmed with a second scan at the next appropriate cycle.
Adverse events (Part 2) | Up to 2 years.
  Evaluate the safety of the combinations According to the National Cancer Institute (NCI) Common Terminology for Adverse Events (CTCAE).
Maximum Plasma Concentration (Cmax) (Part 2) | Up to 2 years.
  the Cmax of 609A in patients with long-term medication.
Area Under the Curve (AUC) (Part 2) | Up to 2 years.
  the AUC of 609A in patients with long-term medication.
Median Progression-free Survival (PFS) (Part 1+2) | Up to 2 years .
  The Kaplan-Meier method will be used to estimate median PFS.
Duration of Response(Part 1+2) | Up to 2 years.
  Duration of response is the mean time to progression for all subjects who responded.
Overall Survival (OS) (Part 1+2) | Up to 2 years .
  The Kaplan-Meier method will be used to estimate median OS.
incidence of anti-609A antibodies(Part 1+2) | Up to 2 years.
  incidence of anti-609A antibodies

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing ji shui tan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No